CLINICAL TRIAL: NCT00646893
Title: Comparison of Embryo Transfer With and Without PGS for the Indication of Advanced Reproductive Age (37-42) in Patients Undergoing ART
Brief Title: Preimplantation Genetic Diagnosis for the Indication of Advanced Reproductive Age
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of appropriate funding
Sponsor: Reprogenetics (Industry)
Responsible Party: Santiago Munne, Reprogenetics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: Reprogenetics-01
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Infertility
Keywords: aneuploidy; miscarriage; pregnancy loss; PGD; PGS; Preimplantation Genetic Diagnosis; chromosome abnormalities; IVF; ART
MeSH Terms: conditions — Infertility; Aneuploidy; Abortion, Spontaneous; Chromosome Aberrations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control: assisted hatching, without Preimplantation Genetic Diagnosis
- 2 (Experimental): Test: embryo biopsy with Preimplantation Genetic Diagnosis
  Interventions: Procedure: Preimplantation Genetic Diagnosis (PGD)

INTERVENTIONS:
Procedure: Preimplantation Genetic Diagnosis (PGD) — one-cell embryo biopsy on day 3 of development. The cell will be analyzed by FISH using probes for X,Y,13,15,16,17,18,21,22 chromosomes. Cells with dubious results will be reanalyzed by "no result rescue" (Colls et al. 2007)
  Other Names: PGS; Preimplantation Genetic Screening
  Arms: 2

SUMMARY:
The objective of this study is to demonstrate that Preimplantation Genetic diagnosis will significantly reduce spontaneous abortions and increase ongoing pregnancy rates in patients of advanced maternal age (37-42) undergoing IVF. We would like to test this hypothesis by a randomized trial performed with the most suitable conditions using very successful IVF laboratories capable to perform the embryo biopsy under strict controlled conditions after proper training and validation of the techniques.

DETAILED DESCRIPTION:
Indications: Patients of advanced reproductive age wishing to receive preimplantation genetic screening in ART.

Objectives: To demonstrate that Preimplantation Genetic diagnosis (PGD) will significantly reduce spontaneous abortions and increase ongoing pregnancy rates in patients of advanced maternal age (37-42) undergoing IVF.

Test Method: Preimplantation Genetic Screening through FISH Treatment: In Vitro Fertilization treatment. The resulting embryos of the test group will undergo embryo biopsy followed by PGD with FISH using a 10-probe test with "no result rescue".

Study Population: 978 infertile women undergoing ART Major Inclusions: Premenopausal infertile women wishing to conceive, aged 37 42 years, inclusive, regular menstrual cycles and screening early follicular phase FSH within normal limits.

Major Exclusions: Clinically significant systemic disease; any contraindication to pregnancy or carrying pregnancy to term; known ASRM Grade III or IV endometriosis; clinically significant abnormal findings on a transvaginal ultrasound within 6 weeks prior to the beginning of OCP treatment; extrauterine pregnancy within 3 months prior to the beginning of OCP treatment; poor response in a previous ART cycle (≤ 3 oocytes retrieved); ≥ 3 prior, initiated, consecutive ART cycles without a clinical pregnancy; prior severe OHSS; TESA and TESE patients; patients carriers of chromosomal or genetic diseases.

Randomization: Eligible patients will be randomized in a 1:1 ratio to either:

Group A: Hatching "or" Group B: Hatching + PGS Study Procedures The study will be conducted on an outpatient basis. All pre-study screening assessments will be performed prior to treatment start.

Post-treatment Oocyte retrieval and embryology procedures will be Procedures performed according to the usual practice of the study center. Test Method Hatching, embryo biopsy, fixation and Fluorescence in-situ Hybridization (FISH) will be performed strictly in line with the methodology included in this protocol and only carried out by technicians certified by Reprogenetics.

Primary Endpoint: ongoing pregnancy rate (past 2nd trimester). Secondary Endpoints: implantation rate, pregnancy rate, miscarriage rate and live birth.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal infertile women wishing to conceive
* Aged 37 42 years, inclusive,
* Regular menstrual cycles (generally 25 35 days in length) and screening early follicular phase FSH within normal limits.

Exclusion Criteria:

* Clinically significant systemic disease;
* Any contraindication to pregnancy or carrying pregnancy to term;
* Known ASRM Grade III or IV endometriosis;
* Clinically significant abnormal findings on a transvaginal ultrasound within 6 weeks prior to the beginning of OCP treatment;
* Extrauterine pregnancy within 3 months prior to the beginning of OCP treatment;
* ≥ 3 prior, initiated, consecutive ART cycles without a clinical pregnancy;
* Prior severe OHSS;
* TESA and TESE patients;
* Patients carriers of chromosomal or genetic diseases.
* Egg donation cycles.
* Frozen Cycles.

Ages: 37 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-01 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy rate (past 2nd trimester). | after 21 days, 20 weeks, and 7 month of treatment

SECONDARY OUTCOMES:
spontaneous abortions | within 1st and 2nd trimester
pregnancy | one month for presence of fetal sac
implantation | first month, for presence of fetal sacs

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Munne, PhD, Principal Investigator — Reprogenetics
Locations (5):
- United States (4):
  - ART Reproductive Center,, Beverly Hills, California
  - Fertility Centers of Illinois, Highland Park, Illinois
  - Institute for Reproductive Medicine and Science at Saint Barnabas Medical Center, Livingston, New Jersey
  - Reprogenetics, Livingston, New Jersey
- IVI Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Colls P, Escudero T, Cekleniak N, Sadowy S, Cohen J, Munne S. Increased efficiency of preimplantation genetic diagnosis for infertility using "no result rescue". Fertil Steril. 2007 Jul;88(1):53-61. doi: 10.1016/j.fertnstert.2006.11.099. Epub 2007 Feb 12. PMID 17296179